CLINICAL TRIAL: NCT01175642
Title: Specificity and Generalizability of Cognitive Remediation and Functional Skills Training in Schizophrenia
Brief Title: Cognitive Remediation and Functional Skills Training in Schizophrenia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Christopher R. Bowie, Professor, National Alliance for Research on Schizophrenia and Depression
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYC-085-08
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2010-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Psychosis; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive remediation (Experimental): Cognitive remediation
  Interventions: Behavioral: Cognitive Remediation
- Functional Adaptive Skills Training (Active Comparator): Functional and social skills group treatment
  Interventions: Behavioral: FAST
- Combined Treatment (Active Comparator): Combined cognitive remediation and functional adaptive skills training
  Interventions: Behavioral: Cognitive Remediation; Behavioral: FAST

INTERVENTIONS:
Behavioral: Cognitive Remediation — Computer-based, therapist-lead cognitive remediation
  Arms: Cognitive remediation; Combined Treatment
Behavioral: FAST — Functional adaptive skills training. Group treatment to foster the acquisition of social and adaptive skills
  Arms: Combined Treatment; Functional Adaptive Skills Training

SUMMARY:
This randomized trial is examining whether a treatment called cognitive remediation is more effective when it is paired with a social and functional skills training component.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Enrolled in outpatient mental health care
* Reading level of 6th grade or higher
* English speaking

Exclusion Criteria:

* Medical conditions known to affect cognition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
neurocognition | 12 weeks

SECONDARY OUTCOMES:
functional competence | 12 weeks
  performance-based measures of functional and social competence
neurocognition | 24 weeks
neurocognition | 36 weeks
functional competence | 24 weeks
functional competence | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Bowie, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowie CR, McGurk SR, Mausbach B, Patterson TL, Harvey PD. Combined cognitive remediation and functional skills training for schizophrenia: effects on cognition, functional competence, and real-world behavior. Am J Psychiatry. 2012 Jul;169(7):710-8. doi: 10.1176/appi.ajp.2012.11091337. PMID 22581070